CLINICAL TRIAL: NCT05587829
Title: Effects of Diaphragm and Abdominal Muscle Training on Pulmonary Function Testing and Dyspnea Among Chronic Obstructive Pulmonary Disease Patients.
Brief Title: Effects of Diaphragm and Abdominal Muscle Training on PFT and Dyspnea Among COPD Obstructive Pulmonary Disease Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aqsa Minahil
Record Dates: First submitted 2022-09-05; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: dyspnea; pulmonary function testing; diaphragmatic training; abdominal training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A: will be treated with basic breathing technique.
  Interventions: Other: basic breathing technique
- Group B (Experimental): Group B: will be treated by will be breathing technique along with diaphragm and abdominal training.
  Interventions: Other: • Diaphragmatic breathing technique; Other: basic breathing technique

INTERVENTIONS:
Other: • Diaphragmatic breathing technique — In supine position, the participant inhales through the mouth for 5 s to expand the abdomen to the maximal level, minimizing movement of the thorax, and performs a long exhalation to maintain a lower abdominal contraction and retroversion of the pelvis
  Other Names: • Abdominal breathing technique
  Arms: Group B
Other: basic breathing technique — Deep Breathing for 15 minutes

SUMMARY:
It will be a randomized control trial at Services Hospital Lahore through convenience sampling technique which will be allocated through simple random sampling through sealed opaque enveloped in to Group A and Group B . Group A: patients will be treated with basic breathing technique whereas Group B: will be treated by will be breathing technique along with diaphragm and abdominal training. The study will be completed within 6 months after synopsis approval from ethical Committee of RCRS & AHS . Data will be entered and analyzed by SPSS version 25. After assessing the normality of data , it will be decided either parametric or non-parametric test will be use within a group or between two groups.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a set of diseases that cause airflow obstruction, breathing difficulties, wheezing and chest tightness. Risk factors are smoking and non-tobacco-smoking, the use of biomass fuel and open fires for domestic purposes in poorly ventilated households. Physiotherapy is an important component of multidisciplinary therapies. Airway clearing, pulmonary rehabilitation, inspiratory muscle training, and non-invasive ventilation is the prior treatment .The aim of this study will be to find the effects of diaphragm and abdominal muscle training on pulmonary function testing and dyspnea among COPD patients .

It will be a randomized control trial at Services Hospital Lahore through convenience sampling technique which will be allocated through simple random sampling through sealed opaque enveloped in to Group A and Group B . Group A: patients will be treated with basic breathing technique whereas Group B: will be treated by will be breathing technique along with diaphragm and abdominal training. The study will be completed within 6 months after synopsis approval from ethical Committee of RCRS & AHS . Data will be entered and analyzed by SPSS version 25. After assessing the normality of data , it will be decided either parametric or non-parametric test will be use within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 35-60 years
* Moderate COPD patients.
* Cognitive
* no previous surgery
* clinically stable COPD patients with reduced inspiratory muscle strength [Pi and persistent activity-related dyspnea

Exclusion Criteria:

* Acute attack
* Severe copd
* Inability to perform physiological testing
* active cardiovascular comorbidity (i.e., severe heart failure with reduced left ventricular ejection fraction, cardiomyopathy, recent acute myocardial infarction, cardiac arrhythmias, or stroke),
* Unstable
* Red Flags Like: Fever, Night Sweats, Malaise

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
• Spirometer for pulmonary function testing FVC | 4 months
  The most effective and common method for diagnosing COPD is spirometry. Its also known as a pulmonary function test or PFT. This easy, painless test measures lung function and capacity. To perform this test, you will exhale as forcefully as possible intoThe most effective and common method for diagnosing COPD is spirometry.
  Its also known as a pulmonary function test or PFT. This easy, painless test measures lung function and capacity. To perform this test, you will exhale as forcefully as possible into a tube connected to the spirometer, a small machine.
  a tube connected to the spirometer, a small machine.
• Spirometer for pulmonary function testing FVC1 | 4 months
  The most effective and common method for diagnosing COPD is spirometry. Its also known as a pulmonary function test or PFT. This easy, painless test measures lung function and capacity. To perform this test, you will exhale as forcefully as possible intoThe most effective and common method for diagnosing COPD is spirometry.
  Its also known as a pulmonary function test or PFT. This easy, painless test measures lung function and capacity. To perform this test, you will exhale as forcefully as possible into a tube connected to the spirometer, a small machine.
  a tube connected to the spirometer, a small machine.

SECONDARY OUTCOMES:
• Dyspnea MDP | 4 months
  Use these scales to rate the intensity of the breathing sensations you feel [felt] (like the loudness of sound, regardless of whether the sensation is pleasant or unpleasant; for example a sensation could be intense without being unpleasant.)

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Zia, PP-DPT, Principal Investigator — Riphah International University

REFERENCES:
- [Background] Olloquequi J. COVID-19 Susceptibility in chronic obstructive pulmonary disease. Eur J Clin Invest. 2020 Oct;50(10):e13382. doi: 10.1111/eci.13382. Epub 2020 Sep 2. PMID 32780415
- [Background] Magitta NF, Walker RW, Apte KK, Shimwela MD, Mwaiselage JD, Sanga AA, Namdeo AK, Madas SJ, Salvi SS. Prevalence, risk factors and clinical correlates of COPD in a rural setting in Tanzania. Eur Respir J. 2018 Jan 31;51(2):1700182. doi: 10.1183/13993003.00182-2017. Print 2018 Feb. PMID 29386343
- [Background] Langer D, Ciavaglia C, Faisal A, Webb KA, Neder JA, Gosselink R, Dacha S, Topalovic M, Ivanova A, O'Donnell DE. Inspiratory muscle training reduces diaphragm activation and dyspnea during exercise in COPD. J Appl Physiol (1985). 2018 Aug 1;125(2):381-392. doi: 10.1152/japplphysiol.01078.2017. Epub 2018 Mar 15. PMID 29543134
- [Background] Waatevik M, Johannessen A, Hardie JA, Bjordal JM, Aukrust P, Bakke PS, Eagan TM. Different COPD disease characteristics are related to different outcomes in the 6-minute walk test. COPD. 2012 Jun;9(3):227-34. doi: 10.3109/15412555.2011.650240. Epub 2012 Apr 12. PMID 22497532
- [Background] Masjedi M, Ainy E, Zayeri F, Paydar R. Assessing the Prevalence and Incidence of Asthma and Chronic Obstructive Pulmonary Disease in the Eastern Mediterranean Region. Turk Thorac J. 2018 Apr;19(2):56-60. doi: 10.5152/TurkThoracJ.2018.17051. Epub 2018 Apr 1. PMID 29755807
- [Background] Ko FW, Chan KP, Hui DS, Goddard JR, Shaw JG, Reid DW, Yang IA. Acute exacerbation of COPD. Respirology. 2016 Oct;21(7):1152-65. doi: 10.1111/resp.12780. Epub 2016 Mar 30. PMID 27028990
- [Background] Yamaguti WP, Claudino RC, Neto AP, Chammas MC, Gomes AC, Salge JM, Moriya HT, Cukier A, Carvalho CR. Diaphragmatic breathing training program improves abdominal motion during natural breathing in patients with chronic obstructive pulmonary disease: a randomized controlled trial. Arch Phys Med Rehabil. 2012 Apr;93(4):571-7. doi: 10.1016/j.apmr.2011.11.026. PMID 22464088
- [Background] Xu W, Li R, Guan L, Wang K, Hu Y, Xu L, Zhou L, Chen R, Chen X. Combination of inspiratory and expiratory muscle training in same respiratory cycle versus different cycles in COPD patients: a randomized trial. Respir Res. 2018 Nov 20;19(1):225. doi: 10.1186/s12931-018-0917-6. PMID 30458805
- [Background] Gosselink R, De Vos J, van den Heuvel SP, Segers J, Decramer M, Kwakkel G. Impact of inspiratory muscle training in patients with COPD: what is the evidence? Eur Respir J. 2011 Feb;37(2):416-25. doi: 10.1183/09031936.00031810. PMID 21282809
- [Background] Lu Y, Li P, Li N, Wang Z, Li J, Liu X, Wu W. Effects of Home-Based Breathing Exercises in Subjects With COPD. Respir Care. 2020 Mar;65(3):377-387. doi: 10.4187/respcare.07121. Epub 2019 Nov 12. PMID 31719191
- [Background] Scherer TA, Spengler CM, Owassapian D, Imhof E, Boutellier U. Respiratory muscle endurance training in chronic obstructive pulmonary disease: impact on exercise capacity, dyspnea, and quality of life. Am J Respir Crit Care Med. 2000 Nov;162(5):1709-14. doi: 10.1164/ajrccm.162.5.9912026. PMID 11069801
- [Background] Bostanci O, Mayda H, Yilmaz C, Kabadayi M, Yilmaz AK, Ozdal M. Inspiratory muscle training improves pulmonary functions and respiratory muscle strength in healthy male smokers. Respir Physiol Neurobiol. 2019 Jun;264:28-32. doi: 10.1016/j.resp.2019.04.001. Epub 2019 Apr 3. PMID 30953791
- [Background] Wang J, Guo S, Zeng M, Yu P, Mo W. Observation of the curative effect of device-guided rehabilitation on respiratory function in stable patients with chronic obstructive pulmonary disease. Medicine (Baltimore). 2019 Feb;98(8):e14034. doi: 10.1097/MD.0000000000014034. PMID 30813125
- [Background] Kim NS, Seo JH, Ko MH, Park SH, Kang SW, Won YH. Respiratory Muscle Strength in Patients With Chronic Obstructive Pulmonary Disease. Ann Rehabil Med. 2017 Aug;41(4):659-666. doi: 10.5535/arm.2017.41.4.659. Epub 2017 Aug 31. PMID 28971051
- [Background] O'Donnell DE, Milne KM, James MD, de Torres JP, Neder JA. Dyspnea in COPD: New Mechanistic Insights and Management Implications. Adv Ther. 2020 Jan;37(1):41-60. doi: 10.1007/s12325-019-01128-9. Epub 2019 Oct 30. PMID 31673990
- [Background] Abdallah SJ, Smith BM, Wilkinson-Maitland C, Li PZ, Bourbeau J, Jensen D. Effect of Abdominal Binding on Diaphragmatic Neuromuscular Efficiency, Exertional Breathlessness, and Exercise Endurance in Chronic Obstructive Pulmonary Disease. Front Physiol. 2018 Nov 14;9:1618. doi: 10.3389/fphys.2018.01618. eCollection 2018. PMID 30487757
- [Background] Leelarungrayub J, Puntumetakul R, Sriboonreung T, Pothasak Y, Klaphajone J. Preliminary study: comparative effects of lung volume therapy between slow and fast deep-breathing techniques on pulmonary function, respiratory muscle strength, oxidative stress, cytokines, 6-minute walking distance, and quality of life in persons with COPD. Int J Chron Obstruct Pulmon Dis. 2018 Dec 5;13:3909-3921. doi: 10.2147/COPD.S181428. eCollection 2018. PMID 30584292
- [Background] Wada JT, Borges-Santos E, Porras DC, Paisani DM, Cukier A, Lunardi AC, Carvalho CR. Effects of aerobic training combined with respiratory muscle stretching on the functional exercise capacity and thoracoabdominal kinematics in patients with COPD: a randomized and controlled trial. Int J Chron Obstruct Pulmon Dis. 2016 Oct 28;11:2691-2700. doi: 10.2147/COPD.S114548. eCollection 2016. PMID 27822031